CLINICAL TRIAL: NCT04367779
Title: PROTONBIOMARKS - Research of Biomarkers of Response to Proton Beam Therapy in Pediatric and Adult Patients: A Genomic, Epigenetic, and Immunological Analysis
Brief Title: Research of Biomarkers of Response to Proton Beam Therapy in Pediatric and Adult Patients.
Acronym: PROTONBIOMARKS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Other Study IDs: ET19-284
Record Dates: First submitted 2020-04-24; First posted 2020-04-29 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Brain Cancer; Meningioma; Sarcoma
Keywords: Proton Beam Therapy; Biomarkers; Pediatric and adult cancers; Proton Therapy
MeSH Terms: conditions — Brain Neoplasms; Meningioma; Sarcoma; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Tumor sample(s) (FFPE and/or Frozen) from primary tumor (biopsy or surgery specimen) Blood sample (only for alive patients) collected at the time of PBT initiation or during any clinical exam performed after validation of inclusion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- A : High Grade Sarcoma: Pediatric and adult patients with High Grade Sarcoma treated or to be treated with Proton Beam Therapy (PBT) and not candidate to surgery before PBT.
- B : Brain tumors: Pediatric and adult patients with Brain Tumors treated or to be treated with Proton Beam Therapy (PBT) and not candidate to surgery before PBT.
- C : Meningioma: Pediatric and adult patients with Meningioma treated or to be treated with Proton Beam Therapy (PBT) and not candidate to surgery before PBT.

SUMMARY:
This trial is a paucicentric, clinico-biological cohort study with retrospective and prospective enrollment, aiming to identify biomarkers predictive of response to Proton Beam Therapy (PBT) in cancer patients (high grade sarcoma, brain tumors and meningioma). This study include collection of clinical data, of tumor samples (collected during standard of care) and a blood sample for alive patients.

DETAILED DESCRIPTION:
The proton beam model policy adopted by the American Society of Radiation Oncology (ASTRO) in 2017 supports proton therapy in primary solid neoplasms in children treated with curative intent. To date, PBT is also recognised in adults as a valid option providing life expectancy > 10 years, for inoperable axial or head and neck sarcomas, low grade brain tumors (i.e. low grade astrocytoma, oligodendroglioma and ependymoma), non-operated meningioma of skull base and other rare clinical situations (re-irradiation, locally aggressive tumor malignant or not arising in sites which preclude R0 or R1 surgical resection). Recently, Jhaveri et al. have reported the retrospective analysis of a National Cancer Data Base (NCDB) and shown an improved overall survival in adult Grade I-IV glioma patients treated with PBT versus patients treated with radiotherapy (XRT). Positive impact on toxicity free survival and general health status of patients were reported in others indications. centers join their expertise (pediatric, brain and sarcoma cancers for Centre Léon Bérard (CLB) and protons for CAL) and their recruitment to optimize the treatment strategy for these patients.

The Centre Leon Bérard recently reported on the ProfilER protocol (NCT01774409). It is the largest molecular characterization program in France with now over 4000 patients included. It enabled to identify genomic biomarkers of radio resistance. In this context, the investigator's proposal is to conduct a genomic, epigenetic, and immunological analysis of patients treated with proton beam therapy with the aim to identify Biomarkers of response to PBT in pediatric and adult patients.

ELIGIBILITY:
Inclusion Criteria:

* I1 Male or female patients, all ages are eligible.
* I2 Confirmed diagnosis of macroscopic tumor previously treated since 2016 (retrospective cohort) or to be treated (prospective cohort) with PBT including one of the following tumor types:Cohort A : high grade sarcoma ; Cohort B: brain tumors; Cohort C: meningioma.
* I3 Presence of at least one measurable lesion before PBT initiation. Post operative situation is possible providing a measurable macroscopic residue, non candidate to a new surgery before PBT.
* I4 Availability of archival representative formalin-fixed, paraffin-embedded (FFPE) and/or frozen tumor sample, with the corresponding hematoxylin and eosin stained slide and a pathological report, meeting the following quality/quantity control (QC) criteria confirmed by a central pathological review: (this sample will be also used to confirm pathological diagnosis ) : at least 20% of tumor cells and a surface area > 5mm2 with > 90μm of depth.
* I5. Performance status before PBT: Lansky Play score for pediatric patients < 12 years of age ≥ 70%; Karnofsky performance status for pediatric patients ≥ 12 years of age ≥ 70%; PS ECOG for adult patients: 0, 1 or 2.
* I6. For prospective cohort : Life-expectancy before PBT > 2 years .
* I7. For prospective cohort : Women of child-bearing potential and men must agree to use (must have used for retrospective cohort) adequate contraception during all the radiotherapy procedure
* I8. For alive patients - Written informed consent from patient, parents if applicable/legal representative, before any study-specific screening procedures, and willingness to comply to study visits and procedures.

Exclusion Criteria:

* E1. Patients previously treated with radiotherapy in the same site (re-irradiation), either with protons or photons
* E2. Pregnant or breast-feeding patients at time of PBT initiation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Alive or Dead cancer patients with high grade sarcoma, brain tumors or meningioma Previously treated with PBT since 2016 (Retrospective cohort) or Patients to be treated with PBT (Prospective cohort)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-09-24 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Identify predictive biomarkers for local response at 6 months after the end of Proton Beam Therapy | At 6 months after the end of Proton Beam Therapy
  Correlation between local tumor response according to RECIST 1.1 criteria and expression of biomarkers defined by using different techniques (HTG, WES, RNAseq, IHC)

SECONDARY OUTCOMES:
To identify predictive biomarkers for clinical outcomes | At 12 months and at 24 months after the end of Proton Beam Therapy
  Correlation between local tumor response according to RECIST 1.1 criteria and expression of biomarkers defined by using different techniques (HTG, WES, RNAseq, IHC)
To identify predictive biomarkers for clinical outcomes | From the start of Proton Beam Therapy until the date of the first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  Correlation between progression free survival and expression of biomarkers expression of biomarkers defined by using different techniques (HTG, WES, RNAseq, IHC)
To identify predictive biomarkers for clinical outcomes | From the start of Proton Beam Therapy until the date of death from any cause, assessed up to 48 months
  Correlation between overall survival and expression of biomarkers defined by using different techniques (HTG, WES, RNAseq, IHC)
To identify predictive biomarkers for clinical outcomes | From the start of Proton Beam Therapy until at least 24 months after the end of Proton Beam Therapy
  Correlation between radiation related toxicity (only Adverse Event (AE) Grade ≥3) according to NCI-CTCAE V5.0. and expression of biomarkers defined by using different techniques (HTG, WES, RNAseq, IHC)

CONTACTS AND LOCATIONS:
Overall Officials: Claude Line, Principal Investigator — Centre Leon Berard
Locations (2):
- France (2):
  - Centre Léon Bérard, Lyon
  - Centre Antoine Lacassagne, Nice